CLINICAL TRIAL: NCT06624475
Title: Randomized Phase II Trial Neoadjuvant Nivolumab + Relatlimab (Opdualag) Versus Nivolumab for Resectable High-Risk Basal Cell Carcinoma
Brief Title: Neoadjuvant Nivolumab + Relatlimab (Opdualag) Versus Nivolumab for Resectable High-Risk Basal Cell Carcinoma
Acronym: NEON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Soo Park, Medical Oncologist, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-1451; 810617 (Other: UCSD Office of IRB Administration (OIA))
Record Dates: First submitted 2024-09-04; First posted 2024-10-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Nivolumab; relatlimab; Opdualag

STUDY DESIGN:
Intervention Model Description: 2:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1 (Experimental): Nivolumab 480 mg intravenous and Relatlimab 160 mg intravenous every 4 weeks, up to 4 cycles.
  Interventions: Drug: Relatlimab plus Nivolumab
- Cohort 2 (Experimental): Nivolumab 480 mg intravenous every 4 weeks, up to 4 cycles.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a fully humanized monoclonal antibody that binds to the Programmed Death-1 (PD-1) receptor, blocking its interactions with Programmed Death-Ligand 1 (PD-L1) and Programmed Death-Ligand 2 (PD-L2), and thus additionally inhibiting PD1-driven immune suppression. Nivolumab: 480 mg via intravenous administration (28 day cycle).
  Other Names: Opdivo
  Arms: Cohort 2
Drug: Relatlimab plus Nivolumab — Relatlimab plus Nivolumab (Opdualag) is supplied as a single dose vial containing 480 mg of Nivolumab and 160 mg Relatlimab for intravenous administration (28 day cycle).
  Other Names: Opdualag
  Arms: Cohort 1

SUMMARY:
This is a Phase 2 clinical trial with a 2:1 randomization comparing neoadjuvant Nivolumab + Relatlimab (Opdualag) vs neoadjuvant Nivolumab in patients with resectable high risk basal cell carcinoma (HR BCC)

DETAILED DESCRIPTION:
Patients will be treated with 4 cycles of neoadjuvant Nivolumab + Relatlimab (Opdualag, cohort 1) or Nivolumab (cohort 2) given every 4 weeks followed by surgical resection. There will be an option to proceed directly to surgery after 2 cycles of therapy should patients have frank progression of disease based on clinical evaluation. There will also be an option to continue with Opdualag or Nivolumab beyond 4 cycles if there is ongoing clinical benefit per investigator discretion. If there is clinical evidence of a clinical complete response, patients may forgo surgery per investigator discretion. The primary outcome of pathologic response rate will be assessed at the time of resection. Patients will then be monitored for disease recurrence and other secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document.
2. Participants must have histologically or cytologically confirmed basal cell carcinoma.
3. Participants must have high risk BCC as defined by size 20 mm or greater in the head and neck region or 40 mm or greater for the trunk/extremities.
4. Participants must have surgically resectable BCC that is at increased risk for cosmetic disfigurement, functional defects, poor oncologic control, or anticipated to require skin grafting or free flap reconstruction per investigator assessment.
5. Participants must have treatment naive BCC.
6. Aged 18 years or older.
7. Eastern Cooperative Oncology Group Performance Status 0 or 1
8. Demonstrates adequate organ function as defined below:

   Adequate bone marrow function
   1. Absolute neutrophil count ≥ 1,500/microliter
   2. Platelets ≥ 100,000/microliter

      Adequate hepatic function
   3. Total bilirubin >1.5 x institutional upper limit of normal (except participants with Glibert Syndrome who must have a total bilirubin level of <3.0xULN)
   4. Aspartate aminotransferase (AST or SGOT) ≤ 3 x institutional upper limit of normal
   5. Alanine transaminase (ALT or SGPT) ≤ 3 x institutional upper limit of normal

      Adequate renal function
   6. Creatinine clearance Calculated creatinine clearance (CrCl) > 30 mL/min (using the Cockcroft Gault formula)
9. Human immunodeficiency virus (HIV) infected individuals on effective anti retroviral therapy with undetectable viral load within 6 months are eligible for this trial. Patients must not have had an AIDS defining opportunistic infection within the last year or a current CD4 count < 350 cells/microliter.
10. For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
11. Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
12. Concurrent malignancy (present during screening) requiring treatment or history o f prior malignancy active within 2 years prior to randomization (i.e., participants with a history of prior malignancy are eligible if treatment was completed at least 2 years before randomization and the patient has no evidence of disease). Participants with history of prior early stage basal/squamous cell skin cancer or non invasive or in situ cancers that have undergone definitive treatment at any time are also eligible.
13. The effects of Opdualag on the on the developing human fetus are unknown. Therefore, the following criteria apply to participants in each study arm:

Cohort 1 Opdualag:

A woman of child bearing potential (WOCBP) is eligible to enroll if using a contraceptive method that is highly effective (with a failure rate of < 1% per year), with low user dependency, during the intervention period and for the duration of treatment with Opdualag plus 5 half lives of study treatment for a total of 5 months post treatment completion and agrees not to donate eggs (ova, oocytes) for the purpose of re production for the same time period.

Cohort 2 nivolumab:

i. Women who are not of childbearing potential are exempt from contraceptive requirements.

ii. Women participants must have documented proof that they are not of childbearing potential.

iii. Women of child bearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study treatment. An extension up to 72 hours prior to the start of study treatment is permissible in situations where results cannot be obtained within the standard 24 hour window. iv. Additional requirements for pregnancy testing during and after study intervention are located in the Schedule of Assessments.

v. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy. vi. WOCBP must agree to follow instructions for method(s) of contraception and as described below and included in the Informed Consent Form.

vii. WOCBP are permitted to use hormonal contraception methods viii. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

1. Is not a WOCBP. OR
2. Is a WOCB P and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency, during the intervention period and for at least 5 months and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction for the same time period.

Exclusion Criteria:

1. Is currently receiving any other investigational agents.
2. Has participated in a study of an investigational product and received study treatment or used an investigational device within 4 weeks of the first dose of study treatment.
3. Hypersensitivity to Opdualag, nivolumab, or any of their excipients.
4. Presence of untreated (symptomatic) central nervous system metastases.
5. Presence of leptomeningeal metastatic disease.
6. Treatment with any live / attenuated vaccine within 30 days of first study treatment.
7. Radiation therapy within 2 weeks prior to first study treatment. Participants must have recovered (i.e., Grade ≤1 or at baseline) from radiation related toxicities prior to first study treatment.
8. Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) within 14 days or other immunosuppressive medications within 30 days of randomization. Note: Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
9. Participants with an active, known, or suspected autoimmune disease. Note: Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
10. Prior allogeneic tissue/solid organ transplant.
11. Severe uncontrolled cardiac disease within 6 months of screening, including but not limited to poorly controlled hypertension , unstable angina, myocardial infarction, congestive heart failure (New York Heart Association Class II or greater), pericarditis within the previous 6 months, cerebrovascular accident, or clinically significant uncontrolled cardiac arrhythmias.
12. Any prior history of myocarditis and/or current diagnosis of myocarditis, regardless of etiology.
13. Troponin T (TnT) or I (TnI) > 2 x institutional upper limit of normal (ULN).

    1. Participants with TnT or TnI levels between > 1× to 2× ULN will be permitted if repeat levels within 24 hours are ≤ 1× ULN. I f TnT or TnI levels are between > 1× to 2× ULN within 24 hours, the participant must be evaluated by a cardiologist. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2× ULN, the participant must be evaluated by a cardiologist.
    2. After cardiologist evaluation, the participant may be considered for randomization if the Investigator assesses a favorable benefit/risk.
14. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study treatment administration or that may interfere with the interpretation of study results and, in the judgement of the investigator, would make the patient an inappropriate candidate for the study.
15. Pregnant women are excluded from this study because Opdualag are immune checkpoint inhibitors with the potential for teratogenic o r abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Opdualag, breastfeeding should be discontinued if the mother is treated prior to initiating study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Pathologic response rate | 2 years
  The primary endpoint of this study is to evaluate the pathologic response rate (pathological complete response [pCR] plus major pathological response [MPR])) and the clinical complete response rate of Opdualag and Nivolumab in patients with resectable High-Risk Basal Cell Carcinoma.
Clinical complete response rate | 2 years
  Clinical complete response rate, per World Health Organization (WHO) Clinical Response Criteria for externally visible tumor(s) which can only be assessed clinically with bidimensional measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Park, MD, Principal Investigator — UC San Diego Health - Moores Cancer Center
Locations (3):
- United States (3):
  - University of California, Irvine, Irvine, California
  - University of California, San Diego Moores Cancer Center, La Jolla, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No